CLINICAL TRIAL: NCT01024621
Title: Comparison of Confocal Laser Endomicroscopy With Standard Endoscopy for the Detection and Evaluation of Gastric Intestinal Metaplasia in a High Risk Population: A Randomized Controlled Trial
Brief Title: Confocal Laser Endomicroscopy for the Detection of Gastric Intestinal Metaplasia: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterolgoy, Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2009SDU-QILU-G06
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Intestinal Metaplasia
Keywords: gastric intestinal metaplasia; Confocal laser endomicroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): confocal laser endomicroscopy
  Interventions: Device: Endomicroscope
- 2 (Active Comparator): standard endoscopy
  Interventions: Device: Standard endoscopy

INTERVENTIONS:
Device: Endomicroscope — Pentax EC3870K, Tokyo, Japan
  Other Names: Pentax EC3870K endomicroscope
  Arms: 1
Device: Standard endoscopy — Pentax EG-2931 gastroscope
  Other Names: Pentax EC2931 gastroscope (Pentax, Tokyo, Japan)
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether confocal laser endomicroscopy can reduce the biopsy number needed per patient for the detection of gastric intestinal metaplasia without the loss of corresponding diagnostic yield.

DETAILED DESCRIPTION:
Gastric intestinal metaplasia is a well-known premalignant lesions for intestinal type gastric cancer. However, present guidelines such as the updated Sydney System require multiple biopsies whereas reveal an unsatisfactory yield considering the detection and surveillance of these lesions. Confocal laser endomicroscopy is a newly developed endoscopic device that enables microscopic view of the digestive tract. Previous study has showed high sensitivity and specificity for in vivo diagnosis of gastric intestinal metaplasia using confocal laser endomicroscopy. This study aims to assess the real number of biopsies that can be reduced for the detection of gastric intestinal metaplasia using confocal laser endomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old ≤ age < 80 years old
* Patients with dyspeptic symptoms and/or with certain risk factors of gastric intestinal metaplasia
* Able to give informed consent.

Exclusion Criteria:

* Esophageal, gastric or duodenal cancer or other malignancy
* Known GIM or intraepithelial neoplasia in upper GI tract
* Scheduled for endoscopic therapy
* History of upper GI tract surgery
* Reflux esophagitis or acute gastritis or peptic ulcers
* Acute upper gastrointestinal bleeding
* Coagulopathy or bleeding disorders
* Allergy to fluorescein sodium
* Pregnant or breast-feeding (for females)
* Impaired renal function

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
the diagnostic yield of gastric intestinal metaplasia | Seven months

SECONDARY OUTCOMES:
the biopsy number needed in each group | Seven months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China